CLINICAL TRIAL: NCT00302445
Title: An Open-Label Pilot Study to Evaluate the Efficacy and Safety of Raptiva (Efalizumab)in Combination With Narrow Band Phototherapy for the Treatment of Moderate to Severe Plaque Psoriasis.
Brief Title: A Safety and Efficacy Study to Evaluate Efalizumab in Combination With UVB for Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: Dermatology Associates, PLLC (Unknown); Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACD3588s
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Efalizumab
Device: Narrow Band Phototherapy

SUMMARY:
An open label, single arm study to evaluate the study and efficacy of efalizumab in combination with NB-UVB. Weeks 1-12 efalizumab will be administered once a week in combination with NB-UVB three times per week. Weeks 13-24 efalizumab monotherapy will continue. Weeks 25-36 subjects will be followed for safety.

Subjects with moderate to severe plaque psoriasis often require more than one therapy to treat their disease. Because of the different mechanisms of action, it is thought that combined efalizumab and NB-UVB may be more effective and have a more rapid onset than either treatment alone.

DETAILED DESCRIPTION:
This is an open label, single arm, phase IV study to evaluate the study and efficacy of efalizumab in combination with NB-UVB. After screening, review of inclusion and exclusion criteria and obtaining informed consent, 20 subjects from two sites (10 subjects per site) will enter the study. The estimated rate of accrual is two subjects per month per site for a total of five months. The estimated date of study conclusion, including follow-up is January 2007.

Weeks 1-12 efalizumab will be administered subcutaneously once a week in combination with NB-UVB three times per week. At week 12, NB-UVB will be discontinued. Weeks 13-24 efalizumab monotherapy will continue to determine whether or not relapse occurs. Relapse is defined as a 50% decrease in total improvement in PASI score from baseline. Weeks 25-36 subjects will be followed for safety. Patients will be transitioned to appropriate treatment at the discretion of the investigator and/or observed closely.

Subjects with moderate to severe plaque psoriasis often require more than one therapy to treat their disease. Because of the different mechanisms of action, it is thought that combined efalizumab and NB-UVB may be more effective (percent subjects who achieve PASI 75 at 12 weeks) and have a more rapid onset than either treatment alone. This study will examine combining efalizumab with NB-UVB phototherapy for twelve weeks. Then, NB-UVB will be discontinued and efalizumab will be continued for an additional twelve weeks to determine if the achieved effect from combination therapy can be sustained with monotherapy.

The follow-up observation period from 25-36 weeks was chosen to permit an adequate amount of time to observe for any signs of disease rebound and/or adverse events after discontinuation of efalizumab and to insure that subjects are treated for such conditions appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given informed consent
* Subject is in generally good health, and an ambulatory male or female adult (18 years or older)
* Subject has moderate to severe plaque psoriasis affecting greater than or equal to 5% body surface area
* Subject is a candidate for efalizumab in combination with narrowband UVB phototherapy in the opinion of the assessing investigator
* If a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception (birth control) for the duration of the study are necessary
* If a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.

Exclusion Criteria:

* Subject is not in generally good health in the opinion of the investigator
* Subject has a history of a phototoxic reaction
* Subject has a history of NB-UVB failure or severe side effects from UVB that resulted in discontinuation of treatment
* Subject has erythrodermic, pustular, inverse or guttate psoriasis
* Subject is currently using other psoriasis treatments
* Subject has used other psoriasis treatments, including herbal products or alternative therapies within 2 months (biologics), 1 month (systemic therapies including methotrexate, cyclosporine and acitretin, PUVA, Broadband UVB, NB-UVB, and tanning beds), or 2 weeks (topical therapies) of first dose of efalizumab or NB-UVB
* Subject is currently enrolled in any other study except non-treatment, biopsy studies
* Subject has a history of any form of cancer, including lymphoma, with the exception of non-melanoma skin cancer
* Subject has a genetic disorder that predisposes to cancer (e.g. xeroderma pigmentosum)
* Subject has a history of squamous cell cancer within the past 5 years or basal cell cancer within the past 3 months in areas that will be treated with NB-UVB
* Subject has a history of significant drug or alcohol abuse
* Pregnant women, nursing mothers, or women planning to become pregnant during the study
* Subject with congenital or acquired immunodeficiency
* Subjects planning to have prolonged exposure to the sun or tanning beds during the study which, in the investigator's clinical judgement, may modify the subject's disease severity
* Subject has a history of lupus erythematosus, bullous pemphigoid or any other photosensitive condition which may worsen with NB-UVB
* Subject is taking a medication that causes photosensitivity at the discretion of the investigator
* Subject has an active infection or sepsis prior history or serious infection or tendency to get infections easily
* Subject has an untreated positive PD
* Subject has a blood disorder, aplastic anemia, bleeding tendency
* Subject is allergic to efalizumab or any of its components
* Subject has any other condition that, in the opinion of the investigator, makes subject a poor candidate for entry into the study
* Subject will be vaccinated with live vaccines (e.g. Flu-Mist) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Percent subjects who reach PASI 75 at week 12. | Week 12

SECONDARY OUTCOMES:
Percent subjects who reach PASI 90 at weeks 12 and 24 | Week 12 and 24
Percent subjects who reach PASI 75 at week 24 | Week 24
Percent subjects who reach PASI 50 at weeks 12 and 24 | Week 12 and 24
Percent subjects who achieve improvement from baseline on | Baseline, Week 12, Week 24
the DLQI at weeks 12 and 24 | Week 12 and Week 24
Percent subjects who relapse between weeks 12 and 24 | Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Leon H Kircik, MD, Principal Investigator — Derm Research, PLLC; Bernard S Goffe, MD, Principal Investigator — Dermatology Associates, PLLC
Locations (2):
- United States (2):
  - Derm Research, PLLC, Louisville, Kentucky
  - Dermatology Associates, PLLC, Seattle, Washington

REFERENCES:
- [Background] Berneburg M, Rocken M, Benedix F. Phototherapy with narrowband vs broadband UVB. Acta Derm Venereol. 2005;85(2):98-108. doi: 10.1080/00015550510025579. PMID 15823900
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Background] Gupta G, Long J, Tillman DM. The efficacy of narrowband ultraviolet B phototherapy in psoriasis using objective and subjective outcome measures. Br J Dermatol. 1999 May;140(5):887-90. doi: 10.1046/j.1365-2133.1999.02820.x. PMID 10354027
- [Background] Ibbotson SH, Bilsland D, Cox NH, Dawe RS, Diffey B, Edwards C, Farr PM, Ferguson J, Hart G, Hawk J, Lloyd J, Martin C, Moseley H, McKenna K, Rhodes LE, Taylor DK; British Association of Dermatologists. An update and guidance on narrowband ultraviolet B phototherapy: a British Photodermatology Group Workshop Report. Br J Dermatol. 2004 Aug;151(2):283-97. doi: 10.1111/j.1365-2133.2004.06128.x. PMID 15327535
- [Background] Weischer M, Blum A, Eberhard F, Rocken M, Berneburg M. No evidence for increased skin cancer risk in psoriasis patients treated with broadband or narrowband UVB phototherapy: a first retrospective study. Acta Derm Venereol. 2004;84(5):370-4. doi: 10.1080/00015550410026948. PMID 15370703
- [Background] Werther WA, Gonzalez TN, O'Connor SJ, McCabe S, Chan B, Hotaling T, Champe M, Fox JA, Jardieu PM, Berman PW, Presta LG. Humanization of an anti-lymphocyte function-associated antigen (LFA)-1 monoclonal antibody and reengineering of the humanized antibody for binding to rhesus LFA-1. J Immunol. 1996 Dec 1;157(11):4986-95. PMID 8943405
- [Background] Fitzpatrick T and Ortonne JP in Fitzpatrick's Dermatology in General Medicine, Editors: Freedberg IM, Eisen AZ, Wolff K, Austen KF, Goldsmith LA, Katz, SI, 6th Edition 2003 McGraw-Hill; Chapter 88, Page 819
- [Background] Sminkels OQ, Prins M, Veeniiuis RT, De Boo T, Gerritsen MJ, Van Der Wilt GJ, Van De Kerkhof PC, Van Der Valk PG. Effectiveness and side effects of UVB-phototherapy, dithranol inpatient therapy and a care instruction programme of short contact dithranol in moderate to severe psoriasis. Eur J Dermatol. 2004 May-Jun;14(3):159-65. PMID 15246941